CLINICAL TRIAL: NCT02193022
Title: A Study for Safety and Efficacy of Miltefosine for Treatment of Children and Adolescents With Post-Kala-azar Dermal Leishmaniasis (PKDL) in Bangladesh and Association of Serum Vitamin E and Exposure to Arsenic With PKDL
Brief Title: Miltefosine for Children With PKDL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-13045
Record Dates: First submitted 2014-06-23; First posted 2014-07-17 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2018-08

CONDITIONS: Post Kala Azar Dermal Leishmaniasis
Keywords: Bangladesh, PKDL, Visceral Leishmaniasis, Children, Miltefosine
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — miltefosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Miltefosine (Experimental)
  Interventions: Drug: Miltefosine

INTERVENTIONS:
Drug: Miltefosine

SUMMARY:
Hypothesis:

Primary hypothesis:

1. Oral treatment with Miltefosine in children with PKDL at allometric daily dose (based on body weight and height) for 12 weeks is safe with a cure rate of ≥95%.

   Secondary hypothesis:
2. Development of PKDL in children and adolescent is genetically predisposed and is associated with IL-10 & IFN-gamma gene polymorphism causing high and low serum level of IL-10 and IFN-gamma respectively.
3. Nutritional & environmental factors such as low serum vitamin E, A, D, Zn & arsenic exposure are associated with PKDL.

DETAILED DESCRIPTION:
Background:

Visceral leishmaniasis also known as kala-azar is a neglected tropical disease affecting the poorest of the poor living in the rural areas of Bangladesh, Nepal, India, South Sudan, Sudan and Brazil with an annual incidence of 500,000 new cases with 10% mortality. Since 2008, the first oral drug Miltefosine (MF) has been introduced for the treatment of VL in Bangladesh, India and Nepal as part of the National VL / Kala-azar (KA) Elimination Program (NKEP) in these three countries. The duration of treatment is 28 days at a dose of 100 mg / day or 50 mg / day for adult with body weight ≥25 KG and< 25 Kg respectively. For children, it is ≤ 2 mg/Kg/24h. The efficacy of MF for VL is 87%, but we have observed that 15% of those develop Post-kala-azar Dermal (PKDL) Leishmaniasis with an annual incidence of about 300 cases, mostly in the Mymensingh district of Bangladesh (the most VL endemic district in the country). The clinical manifestation of PKDL is macular/papular/nodular /mixed lesions. Children and adolescents with PKDL are otherwise clinically healthy, but these patients continue to carry the parasites for years and can transmit the parasites to others through sand fly bite. In this way these patients play a role as inter-epidemic reservoirs and can initiate new outbreaks of VL in the community. The only current treatment option is 120 injections with SSG (one injection per day for 20 consecutive days in a month for 6 months). Injections are very painful and associated with risks including sudden heart failure from cardiac arrhythmias and death. Therefore, PKDL patients usually do not seek treatment and the compliance is very low, when they take treatment with SSG. Thus, a safe and effective treatment which can ensure better compliance is urgently needed. Recent studies in India showed that 12 weeks treatment with MF of adult PKDL patients is effective (94%) and safe. However, the study reported only 24 adult PKDL cases. Similar results have been observing with adult PKDL patients in Nepal. There is no information about the safety and efficacy of 12 weeks MF treatment of children with PKDL and about pharmacokinetics of MF among these children. It is established that exposure to MF in VL children was less to oral MF at conventional dose of 2.5mg/Kg/day, thus allometric dosing of MF is now recommended by experts. A study is therefore urgently needed for efficacy and safety of allometric daily dose of MF for 12 weeks for treatment of PKDL in children.

Risk factors for PKDL are poorly investigated. Younger age of VL patients and genetic susceptibility to PKDL are found to contribute to PKDL. Exposure to arsenic through drinking water and protein-energy malnutrition are public health problem in Bangladesh. Both arsenic and vitamin E and other nutrients deficiency may contribute to PKDL directly or in combination, because they inhibit innate and adaptive immunity to infections.

Hypothesis(es) and Aims:

1. Oral treatment with Miltefosine in children with PKDL at allometric daily dose for 12 weeks is safe with a cure rate of ≥95%; 2. Development of PKDL in children and adolescent is genetically predisposed and is associated with IL-10 & IFN-gamma gene polymorphism causing high serum level of IL-10 and low serum level of IFN-gamma; 3. Nutritional & environmental factors such as low serum vitamin E & arsenic exposure are associated with PKDL .

Study design:

The study includes a cross sectional survey for suspected PKDL patients among children treated for VL in the past, followed by an open clinical trial with MF with 12 months follow up after treatment and a simultaneous case-control study for PKDL risk factors. Parasitologically confirmed (demonstration of parasite in skin specimens by microscopy and / qPCR) PKDL children will be subjects of the open clinical trial with oral Miltefosine (MF) at allometric daily dose. In the case-control component of the study, confirmed PKDL children will be cases. Children treated for VL in the past and currently without skin lesions will be the controls and will be matched with cases by geographic area, age, sex and time of VL treatment. Inclusion criteria are: a child treated for VL in the past, aged more than 2 years old and less than 18 years old, either sex, fulfill case definition as PKDL case / control, parents / guardian consent for participation of the child in the study. Exclusion criteria are: do not fulfill all inclusion criteria for a case/control, with skin fungal infection / leprosy, without clinical evidence for arsenic dermatosis, negative for rK39 rapid test, control child who will develop PKDL during follow up. Based on expected 95% cure rate, a sample size of 73 PKDL children would produce a two-sided 95% confidence interval with an estimated precision of 5%. Allowing for an attrition rate of 10%, the final sample size is 80 children in each group and the total sample size is 160. Blood, urine and hair specimens will be collected from cases before treatment and at 12 months follow up, and from controls at baseline only. Primary outcome is safety and cure rate of 12 weeks treatment with MF. Cure will be defined by resolution of skin lesions by ≥90% and skin and blood specimens negative for LD bodies and leishmania DNA at 12 months after treatment. Safety will be measured by frequency of adverse events (AEs). We expect transient AEs like vomiting and diarrhea in less than 30% and serious adverse event in none.

Potential Impact:

If 12 weeks treatment with MF at allometric daily dose is found safe and effective for treatment in children with PKDL, then it will be scale up through the National VL Elimination Program. Through the case-control component, we may find nutritional / environmental risk factor for PKDL which will help to design preventative strategy against PKDL.

ELIGIBILITY:
Inclusion Criteria:

* a child of either sex, treated for VL in the past, currently with skin lesions like PKDL, positive for rK39 test, and positive for Leishmania LD bodies by microscopy and / DNA by qPCR in their skin specimens
* more than 2 years and less than 18 years old
* clinically healthy and free from other chronic illness
* received no treatment for PKDL in the last 6 months
* normal hepatic, renal, and hematological functions
* parent / guardian provided informed voluntary written consent for his/her child participation

Exclusion Criteria:

* do not fulfill inclusion criteria
* lesions with mucosal involvement
* serious concomitant illness
* cannot be followed up

Ages: 730 Days to 6569 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
1. Safety of 12 weeks treatment with Miltefosine at allometric dose in children ages < 18 years old. | 15 months
  Safety will be measured by the frequency of the adverse events.
2. Cure rate of 12 weeks treatment with Miltefosine at allometric dose in children ages < 18 years old. | 15 months
  Cure will be defined by the resolution of skin lesion by ≥ 90% and skin and blood specimens negative for leishmania donovani bodies and leishmania DNA at 12 months after treatment.

OTHER OUTCOMES:
Find out the genetic susceptibility to PKDL through evaluation of the association of PKDL development with IL-10 and INF-gamma gene polymorphism. | 15 months
  This will be measured by the association by PKDL and above mentioned genetic polymorphism. Here matched children who will be found during cross sectional survey for PKDL suspects will serve as controls.
Find out the association of developing PKDL with host nutritional factor such as vitamin E, A, D and Zn status and exposure to environmental toxin such as arsenic. | 15 months
  This will be measured by investigating the association of each of these nutritional factors and arsenic with the development of PKDL where matched children without PKDL will serve as control.

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrheal Disease Research, Bangladesh, Dhaka, Bangladesh

REFERENCES:
- [Background] Chrusciak-Talhari A, Dietze R, Chrusciak Talhari C, da Silva RM, Gadelha Yamashita EP, de Oliveira Penna G, Lima Machado PR, Talhari S. Randomized controlled clinical trial to access efficacy and safety of miltefosine in the treatment of cutaneous leishmaniasis Caused by Leishmania (Viannia) guyanensis in Manaus, Brazil. Am J Trop Med Hyg. 2011 Feb;84(2):255-60. doi: 10.4269/ajtmh.2011.10-0155. PMID 21292895
- [Derived] Mondal D, Hasnain MG, Hossain MS, Ghosh D, Ghosh P, Hossain H, Baker J, Nath R, Haque R, Matlashewski G, Hamano S. Study on the safety and efficacy of miltefosine for the treatment of children and adolescents with post-kala-azar dermal leishmaniasis in Bangladesh, and an association of serum vitamin E and exposure to arsenic with post-kala-azar dermal leishmaniasis: an open clinical trial and case-control study protocol. BMJ Open. 2016 May 17;6(5):e010050. doi: 10.1136/bmjopen-2015-010050. PMID 27188804